CLINICAL TRIAL: NCT01690520
Title: Multi-Center, Open-Label Randomized Study of Single or Double Myeloablative Cord Blood Transplantation With or Without Infusion of Off-The-Shelf Ex Vivo Expanded Cryopreserved Cord Blood Progenitor Cells in Patients With Hematologic Malignancies
Brief Title: Donor Umbilical Cord Blood Transplant With or Without Ex-vivo Expanded Cord Blood Progenitor Cells in Treating Patients With Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, Chronic Myelogenous Leukemia, or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nohla Therapeutics, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2603.00; NCI-2012-01572 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2603; 2603.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); P50HL110787 (NIH)
Record Dates: First submitted 2012-09-19; First posted 2012-09-21 (Estimated); Results first posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Acute Biphenotypic Leukemia; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes | interventions — Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Thiotepa; Whole-Body Irradiation; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (standard of care) (Active Comparator): CONDITIONING REGIMEN: One of two possible conditioning regimens is chosen by the attending physician: Patients receive fludarabine phosphate IV over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 to -6., and undergo high dose TBI BID on days -4 to -1 OR Patients receive fludarabine phosphate IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 4 hours on days -5 to -4, and undergo middle intensity TBI QD on days -2 to -1.
  TRANSPLANT: Patients undergo single-unit or double-unit unmanipulated UCB transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclosporine IV over 1 hour BID (adults) or TID (children) or PO on days -3 to 100 with taper beginning on day 101. Patients also receive MMF IV TID a day on days 0-7 then may receive MMF PO TID. Patients remain on MMF TID for a minimum of 30 days, and then may begin a taper if there is no evidence of GVHD and are well-engrafted from one donor unit.
  Interventions: Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Drug: Mycophenolate Mofetil; Drug: Thiotepa; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation
- Arm II (experimental) (Experimental): CONDITIONING REGIMEN: Patients receive the conditioning regimen chosen by the attending physician as in Standard of Care Arm.
  TRANSPLANT: Patients undergo single-unit or double-unit unmanipulated UCB transplant on day 0. Patients also undergo infusion of ex vivo-expanded cord blood progenitor cell infusion at least 4 hours after completion of UCB transplant.
  GVHD PROPHYLAXIS: Patients receive cyclosporine IV or PO and mycophenolate mofetil IV or PO as in Standard of Care Arm.
  Interventions: Drug: Cyclophosphamide; Drug: Cyclosporine; Biological: Ex Vivo-Expanded Cord Blood Progenitor Cell Infusion; Drug: Fludarabine Phosphate; Drug: Mycophenolate Mofetil; Drug: Thiotepa; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
Drug: Cyclosporine — Given IV or PO
Biological: Ex Vivo-Expanded Cord Blood Progenitor Cell Infusion — Given IV
  Other Names: NLA101; Dilanubicel
  Arms: Arm II (experimental)
Drug: Fludarabine Phosphate — Given IV
Drug: Mycophenolate Mofetil — Given IV or PO
Drug: Thiotepa — Given IV
Radiation: Total-Body Irradiation — Undergo high dose or middle intensity TBI
Procedure: Umbilical Cord Blood Transplantation — Undergo single-unit or double-unit unmanipulated umbilical cord blood transplant
  Other Names: Cord Blood Transplantation; UCB transplantation

SUMMARY:
This randomized phase II trial studies how well donor umbilical cord blood transplant with or without ex-vivo expanded cord blood progenitor cells works in treating patients with acute myeloid leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, or myelodysplastic syndromes. Giving chemotherapy and total-body irradiation before a donor umbilical cord blood transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's cells. When the healthy stem cells and ex-vivo expanded cord blood progenitor cells are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. It is not yet known whether giving donor umbilical cord blood transplant plus ex-vivo expanded cord blood progenitor cells is more effective than giving a donor umbilical cord blood transplant alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the time to neutrophil engraftment (absolute neutrophil count [ANC] >= 500) in patients receiving a standard of care myeloablative cord blood transplant (CBT) augmented with an off-the-shelf pre-expanded and cryopreserved cord blood product to those who do not receive the product.

SECONDARY OBJECTIVES:

I. Provide initial data on clinical and economic benefit, such as time to platelet engraftment, duration of initial hospitalization, transplant-related mortality (TRM), death without engraftment, and incidence of severe infections in the first 100 days post-transplant.

II. The kinetics of immune system recovery will also be evaluated in both arms.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Standard of Care Arm:

CONDITIONING REGIMEN: One of two possible conditioning regimens is chosen by the attending physician: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 to -6., and undergo high dose total-body irradiation (TBI) twice daily (BID) on days -4 to -1 OR, patients receive fludarabine phosphate IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 4 hours on days -5 to -4, and undergo middle intensity TBI once daily (QD) on days -2 to -1.

TRANSPLANT: Patients undergo single-unit or double-unit unmanipulated umbilical cord blood (UCB) transplant on day 0.

GRAFT-VERSUS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients receive cyclosporine IV over 1 hour BID (adults) or thrice daily (TID) (children) or orally (PO) on days -3 to 100 with taper beginning on day 101. Patients also receive mycophenolate mofetil (MMF) IV TID on days 0-7 then may receive MMF PO TID. Patients remain on MMF TID for a minimum of 30 days, and then may begin taper if there is no evidence of GVHD and are well-engrafted from one donor unit.

Experimental Arm:

CONDITIONING REGIMEN: Patients receive the conditioning regimen chosen by the attending physician as in Standard of Care Arm.

TRANSPLANT: Patients undergo single-unit or double-unit unmanipulated UCB transplant on day 0. Patients also receive an infusion of ex vivo-expanded cord blood progenitors at least 4 hours after completion of UCB transplant.

GVHD PROPHYLAXIS: Patients receive cyclosporine IV or PO and mycophenolate mofetil IV or PO as in Standard of Care Arm.

After completion of study treatment, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age criteria:

  * High dose TBI regimen: 6 months to =< 45 years
  * Middle intensity TBI regimen: 6 months to =< 65 years
  * Conditioning regimen selection should be based on the underlying disease, presence of minimal residual disease (MRD), age, co-morbidities, attending physician, and site preference; conditioning regimen will not require stratification of the randomization due to heterogeneity in the cohort of eligible patients.
* Acute myeloid leukemia, including biphenotypic acute leukemia or mixed-lineage leukemia

  * All patients must have acute myeloid leukemia (AML) that is considered best treated by stem cell transplant by the referring physician and the attending transplant physician
  * All patients must be in complete remission (CR) as defined by < 5% blasts by morphology/flow cytometry in a representative bone marrow sample with cellularity >= 15% for age
  * Patients in which adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry, recovery of peripheral blood counts with no circulating blasts, and/or normal cytogenetics (if applicable) may still be eligible; reasonable attempts must be made to obtain an adequate specimen for morphologic assessment, including possible repeat procedures; these patients must be discussed with the principal investigator prior to enrollment
* Acute lymphoblastic leukemia, including biphenotypic acute leukemia or mixed-lineage leukemia

  * High risk first complete remission (CR1) (for example, but not limited to: t(9;22), t(1;19), t(4;11) or other mixed-lineage leukemia [MLL] rearrangements, hypodiploid); or high risk (HR) as defined by referring institution treatment protocol greater than 1 cycle to obtain CR; second complete remission (CR2) or greater
  * All patients must be in CR as defined by < 5% blasts by morphology/flow cytometry in a representative bone marrow sample with cellularity >= 15% for age
  * Patients in which adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry, recovery of peripheral blood counts with no circulating blasts, and/or normal cytogenetics (if applicable) may still be eligible; reasonable attempts must be made to obtain an adequate specimen for morphologic assessment, including possible repeat procedures; these patients must be discussed with the principal investigator prior to enrollment
* Chronic myelogenous leukemia excluding refractory blast crisis; to be eligible in first chronic phase (CP1) patient must have failed or be intolerant to tyrosine kinase inhibitor therapy
* Myelodysplasia (MDS) International Prognostic Scoring System (IPSS) intermediate (Int)-2 or high risk (i.e., refractory anemia with excess blasts [RAEB], refractory anemia with excess blasts in transformation [RAEBt]) or refractory anemia with severe pancytopenia or high risk cytogenetics; blasts must be < 10% by a representative bone marrow aspirate morphology
* Karnofsky (>= 16 years old) >= 70 or Eastern Cooperative Oncology Group (ECOG) 0-1
* Lansky (< 16 years old) >= 60
* Adults: calculated creatinine clearance must be > 60 mL and serum creatinine =< 2 mg/dL
* Children (< 18 years old): calculated creatinine clearance must be > 60 mL/min
* Total serum bilirubin must be < 3 mg/dL unless the elevation is thought to be due to Gilbert's disease or hemolysis
* Transaminases must be < 3 x the upper limit of normal per reference values of referring institution
* Diffusing capacity of the lung for carbon monoxide (DLCO) corrected > 60% normal
* For pediatric patients unable to perform pulmonary function tests, oxygen (O2) saturation > 92% on room air
* May not be on supplemental oxygen
* Left ventricular ejection fraction > 45% OR
* Shortening fraction > 26%
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Uncontrolled viral or bacterial infection at the time of study enrollment
* Active or recent (prior 6 month) invasive fungal infection without infectious disease (ID) consult and approval
* History of human immunodeficiency virus (HIV) infection
* Pregnant or breastfeeding
* Prior myeloablative transplant containing full dose TBI (greater than 8 Gy)
* Central nervous system (CNS) leukemic involvement not clearing with intrathecal chemotherapy and/or cranial radiation prior to initiation of conditioning; diagnostic lumbar puncture is to be performed per protocol
* Patients >= 45 years: comorbidity score of 5 or higher

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Milano, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (8):
- United States (8):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of Colorado, Denver, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Full Analysis Set includes all randomized subjects (78 in Arm I SOC and 82 in Arm II Expanded Arm). The modified intent to treat (mITT) analysis set requires subjects in the FAS to undergo hematopoietic cell transplant (HCT) and receive study drug. Two subjects in Arm II withdrew prior to receiving study drug and are therefore not included in the mITT analysis set (78 in SOC and 80 in Expanded Arm).
Groups:
- Arm I (Standard of Care): CONDITIONING REGIMEN: One of two possible conditioning regimens is chosen by the attending physician: Patients receive fludarabine phosphate IV over 30 minutes on days -8 to -6, cyclophosphamide IV on days -7 to -6., and undergo high dose TBI BID on days -4 to -1 OR Patients receive fludarabine phosphate IV over 30-60 minutes on days -6 to -2, cyclophosphamide IV on day -6, thiotepa IV over 4 hours on days -5 to -4, and undergo middle intensity TBI QD on days -2 to -1.
  TRANSPLANT: Patients undergo single-unit or double-unit unmanipulated UCB transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclosporine IV over 1 hour BID (adults) or TID (children) or PO on days -3 to 100 with taper beginning on day 101. Patients also receive MMF IV TID a day on days 0-7 then may receive MMF PO TID. Patients remain on MMF TID for a minimum of 30 days, and then may begin a taper if there is no evidence of GVHD and are well-engrafted from one donor unit.
  Cyclophosphamide: Given IV
  Cyclosporine: Given IV or PO
  Fludarabine Phosphate: Given IV
  Mycophenolate Mofetil: Given IV or PO
  Thiotepa: Given IV
  Total-Body Irradiation: Undergo high dose or middle intensity TBI
  Umbilical Cord Blood Transplantation: Undergo single-unit or double-unit unmanipulated umbilical cord blood transplant
- Arm II (Experimental): CONDITIONING REGIMEN: Patients receive the conditioning regimen chosen by the attending physician as in Standard of Care Arm.
  TRANSPLANT: Patients undergo single-unit or double-unit unmanipulated UCB transplant on day 0. Patients also undergo infusion of ex vivo-expanded cord blood progenitor cell infusion at least 4 hours after completion of UCB transplant.
  GVHD PROPHYLAXIS: Patients receive cyclosporine IV or PO and mycophenolate mofetil IV or PO as in Standard of Care Arm.
  Cyclophosphamide: Given IV
  Cyclosporine: Given IV or PO
  Ex Vivo-Expanded Cord Blood Progenitor Cell Infusion: Given IV
  Fludarabine Phosphate: Given IV
  Mycophenolate Mofetil: Given IV or PO
  Thiotepa: Given IV
  Total-Body Irradiation: Undergo high dose or middle intensity TBI
  Umbilical Cord Blood Transplantation: Undergo single-unit or double-unit unmanipulated umbilical cord blood transplant
Period: Overall Study
Arm/Group | Arm I (Standard of Care) | Arm II (Experimental)
Started | 78 | 82
Modified Intent to Treat (mITT) | 78 | 80
Completed | 27 | 35
Not Completed | 51 | 47
Not completed — Death | 25 | 21
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Relapse | 0 | 1
Not completed — Other | 0 | 1
Not completed — Ongoing Follow-Up at time of Analysis | 22 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Standard of Care) | Arm II (Experimental) | Total
Number analyzed (Participants) | 78 | 82 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 24 | 51
  Between 18 and 65 years | 51 | 58 | 109
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.76 (14.858) | 27.72 (14.699) | 27.25 (14.738)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 40 | 67
  Male | 51 | 42 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 18 | 37
  Not Hispanic or Latino | 59 | 57 | 116
  Unknown or Not Reported | 0 | 7 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 15 | 10 | 25
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 6 | 4 | 10
  White | 34 | 52 | 86
  More than one race | 7 | 9 | 16
  Unknown or Not Reported | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 78 | 82 | 160
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 160.09 (23.481) | 159.85 (24.680) | 159.97 (24.028)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 67.70 (26.886) | 69.77 (27.103) | 68.76 (26.933)
Cord Blood Units Received [Count of Participants; unit: Participants]
  1 Cord Blood Unit | 22 | 17 | 39
  2 Cord Blood Units | 56 | 65 | 121

OUTCOME MEASURES:

1. Primary Outcome: Time to Neutrophil Engraftment
Description: First of two consecutive days with absolute neutrophil count (ANC) equal to or greater than 500 cell/microliter measured from day of transplant.
Time Frame: Up to 55 days post-transplant
Population: The primary analysis set for the analysis of Neutrophil Enrgraftment and Platelet Engraftment was the modified intent to treat (mITT) analysis set. The difference between the full analysis set (FAS) and the mITT is the requirement to undergo hematopoietic cell transplant (HCT) and receive study drug. Two subjects in Arm II withdrew prior to receiving study drug, and are therefore not included in the mITT analysis set, nor the primary efficacy analyses.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm I (Standard of Care) | Arm II (Experimental)
Number analyzed (Participants) | 72 | 75
days | 20.0 [19.0 to 22.0] | 22.0 [20.0 to 24.0]

2. Secondary Outcome: Time to Platelet Engraftment (20k)
Description: First day of seven consecutive days with platelet count equal to or greater than 20,000 cells/microliter without platelet transfusions measured from day of transplant.
Time Frame: Up to 100 days post-transplant
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm I (Standard of Care) | Arm II (Experimental)
Number analyzed (Participants) | 65 | 66
days | 40.0 [34.0 to 42.0] | 38.0 [35.0 to 43.0]

3. Secondary Outcome: Overall Survival
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Standard of Care) | Arm II (Experimental)
Number analyzed (Participants) | 78 | 80
Participants | 52 | 57

4. Secondary Outcome: Non-relapse Mortality
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Standard of Care) | Arm II (Experimental)
Number analyzed (Participants) | 78 | 80
Participants | 16 | 16

5. Secondary Outcome: Proportion of Patients With Severe Acute Graft Versus Host Disease
Time Frame: Up to 100 days post-transplant
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Standard of Care) | Arm II (Experimental)
Number analyzed (Participants) | 78 | 80
proportion of participants | 0.14 [0.07 to 0.24] | 0.16 [0.09 to 0.26]

6. Secondary Outcome: Proportion of Participants With Chronic Graft Versus Host Disease
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Standard of Care) | Arm II (Experimental)
Number analyzed (Participants) | 78 | 80
Participants | 27 | 23

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | Arm I (Standard of Care) | Arm II (Experimental)
All-Cause Mortality (participants affected / at risk) | 25/78 | 21/82
Serious Adverse Events (participants affected / at risk) | 48/78 | 55/82
Other Adverse Events (participants affected / at risk) | 71/78 | 73/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Standard of Care) (N=78) | Arm II (Experimental) (N=82)
Pyrexia (General disorders) | 14 | 17
Multiple organ dysfunction syndrome (General disorders) | 1 | 2
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Complication associated with device (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus gastritis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Oral infection (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 5
Staphylococcal infection (Infections and infestations) | 2 | 2
BK virus infection (Infections and infestations) | 1 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 2 | 0
Pneumonia fungal (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Jejunal perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Colitis (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3
Acute graft versus host disease in intestine (Immune system disorders) | 1 | 2
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Acute graft versus host disease in liver (Immune system disorders) | 1 | 1
Graft versus host disease (Immune system disorders) | 5 | 7
Haematuria (Renal and urinary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 4
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3
Transplant failure (Injury, poisoning and procedural complications) | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Lymphatic disorder (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Standard of Care) (N=78) | Arm II (Experimental) (N=82)
Decreased appetite (Metabolism and nutrition disorders) | 39 | 38
Hypokalemia (Metabolism and nutrition disorders) | 14 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1
Iron overload (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 7 | 9
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 2 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 30 | 36
Nausea (Gastrointestinal disorders) | 15 | 25
Diarrhoea (Gastrointestinal disorders) | 11 | 11
Vomiting (Gastrointestinal disorders) | 5 | 9
Abdominal pain (Gastrointestinal disorders) | 8 | 4
Embolism (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 43 | 42
Hypotension (Vascular disorders) | 7 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 37 | 40
Rash (Skin and subcutaneous tissue disorders) | 3 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Enterococcal infection (Infections and infestations) | 5 | 3
Adenovirus infection (Infections and infestations) | 4 | 2
Alpha haemolytic streptococcal infection (Infections and infestations) | 5 | 1
Cystitis (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 3 | 3
BK virus infection (Infections and infestations) | 1 | 3
Device related infection (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 1 | 3
Candida infection (Infections and infestations) | 2 | 0
Encephalitis (Infections and infestations) | 0 | 2
Escherichia infection (Infections and infestations) | 1 | 1
Human polyomavirus infection (Infections and infestations) | 2 | 0
Pseudomonas infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Stomatococcal infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Actinomycotic sepsis (Infections and infestations) | 1 | 0
Administration site cellulitis (Infections and infestations) | 1 | 0
Bacillus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Coronavirus infection (Infections and infestations) | 1 | 0
Corynebacterium infection (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 1 | 0
Enterocolitis infection (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Fusobacterium infection (Infections and infestations) | 0 | 1
Gastric infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Leuconostoc infection (Infections and infestations) | 0 | 1
Lip infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 7 | 5
Lung infection (Infections and infestations) | 7 | 6
Human herpesvirus 6 infection (Infections and infestations) | 6 | 5
Cytomegalovirus infection (Infections and infestations) | 2 | 7
Streptococcal infection (Infections and infestations) | 7 | 2
Bacterial infection (Infections and infestations) | 4 | 1
Clostridium difficile infection (Infections and infestations) | 3 | 0
Blood bilirubin increased (Investigations) | 11 | 8
Alanine aminotransferase increased (Investigations) | 3 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 2
Blood aluminium increased (Investigations) | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Weight decreased (Investigations) | 2 | 0
White blood cell count increased (Investigations) | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Urine output decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 13 | 9
Neutrophil count decreased (Investigations) | 8 | 3
White blood cell count decreased (Investigations) | 4 | 1
Blood creatinine increased (Investigations) | 1 | 6
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Seizure (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 9 | 5
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 1 | 2
Fatigue (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pneumatosis (General disorders) | 1 | 0
Pain (Gastrointestinal disorders) | 8 | 3
Pyrexia (Gastrointestinal disorders) | 1 | 2
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 5 | 4
Depression (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Pericardial effusion (Cardiac disorders) | 2 | 2
Cardiac failure (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 2
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT01690520/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT01690520/SAP_001.pdf